CLINICAL TRIAL: NCT02804451
Title: Intubation During Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03/02/2016
Record Dates: First submitted 2016-06-11; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Endotracheal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation without chest compression (Experimental): normal airway, without chest compression during intubation.
  Interventions: Device: Macintosh laryngoscope; Device: TruView EVO2 laryngoscope; Device: TruView EVO2 PCD laryngoscope; Device: ETView SL
- Intubation with uninterrupted chest compression (Experimental): normal airway, with continuous chest compressions
  Interventions: Device: Macintosh laryngoscope; Device: TruView EVO2 laryngoscope; Device: TruView EVO2 PCD laryngoscope; Device: ETView SL

INTERVENTIONS:
Device: Macintosh laryngoscope — intubation with standard macintosh larygoscope; gold standard
  Other Names: MAC
Device: TruView EVO2 laryngoscope — A TruView EVO2 laryngoscope with blade size 3 (EVO2; Truphatek Holdings, Ltd., Netanya, Israel),
  Other Names: EVO2
Device: TruView EVO2 PCD laryngoscope — A TruView EVO2 PCD laryngoscope with blade size 3 (PCD; Truphatek Interbational Ltd., Netanya, Israel),
  Other Names: PCD
Device: ETView SL — An ETView SL (ETView; ETViewLtd, Misgav, Israel) ednotracheal tube
  Other Names: ETView

SUMMARY:
The aim of the study was to compare the intubation time and effectiveness, the grade of larynx visibility, and the ease of intubation in adults performed by nurses using 4 devices: a Macintosh blade laryngoscope (MAC), and a TruView EVO2 (EVO2), TruView EVO2 PCD (PCD), and ETView SL (ETView) laryngoscope, in simulated CPR settings with and without CC.

ELIGIBILITY:
Inclusion Criteria:

* had not received any training in endotracheal intubation with videolaryngoscopy before the study,
* had nursing specialization in anaesthesiology or emergency medicine,
* presented with no wrist or low back diseases or pregnancy.

Exclusion Criteria:

* not meet the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
time to the first ventilation attempt | 1 day

SECONDARY OUTCOMES:
time to visualize the larynx | 1 day
time to introduce the endotracheal tube through the vocal cords | 1 day
success rate | 1 day
  first intubation attempt success rate
degree of larynx visibility | 1 day
  analysed based on a Cormack-Lehane scale
ease of intubation technique | 1 day
  10-point visual analogue scale (VAS) was used, where 1 indicated an extremely simple procedure, while 10 - an extremely difficult one

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

REFERENCES:
- [Background] Kurowski A, Szarpak L, Truszewski Z, Czyzewski L. Can the ETView VivaSight SL Rival Conventional Intubation Using the Macintosh Laryngoscope During Adult Resuscitation by Novice Physicians?: A Randomized Crossover Manikin Study. Medicine (Baltimore). 2015 May;94(21):e850. doi: 10.1097/MD.0000000000000850. PMID 26020389